CLINICAL TRIAL: NCT01524341
Title: A Proof-of-concept, Open Label, 3-day Repeated Dose Study to Assess Efficacy, Safety, Tolerability and Pharmacokinetics of KAE609 in Adult Patients With Acute, Uncomplicated Plasmodium Falciparum or Vivax Malaria Mono-infection
Brief Title: Efficacy, Safety, Tolerability and Pharmacokinetics of KAE609 in Adult Patients With Acute, Uncomplicated Plasmodium Falciparum or Vivax Malaria Mono-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKAE609X2201
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Malaria
Keywords: Acute malaria; KAE609
MeSH Terms: conditions — Malaria; Acute malaria | interventions — NITD 609

ARMS (2):
- Cohort 1 (Experimental): 10 subjects with Plasmodium vivax malaria will receive 30 mg KAE609 once a day for three days
  Interventions: Drug: KAE609
- Cohort 2 (Experimental): 10 subjects with Plasmodium falciparum malaria will receive 30 mg KAE609 once a day for three days
  Interventions: Drug: KAE609

INTERVENTIONS:
Drug: KAE609 — KAE609 was supplied as capsules for oral use.

SUMMARY:
This study will assess efficacy, safety , tolerability and PK in uncomplicated adult malaria patients with P. vivax or P. falciparum infection after 3 day dosing with KAE609 at 30 mg/day

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 20 to 60 years
* Presence of mono-infection of P. falciparum or P. vivax
* Weight between 40 kg to 90 kg

Exclusion Criteria:

* Patients with signs and symptoms of severe/complicated malaria
* Mixed Plasmodium infection
* Presence of other serious or chronic clinical condition requiring hospitalization.
* Severe malnutrition
* Significant chronic medical conditions which in the opinion of the investigator preclude enrollment into the study

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Parasite clearance time | From baseline to the time point when the blood parasite count is zero(up to a maximum of 5 days)
  Calculated based on parasite count in blood. In thin film, use actual WBCs/µl, of blood to calculate parasite density by using the following formula: parasites/µl= #parasites× actual WBC/#WBCs counted. In thick film, assume that there are 250 RBCs per HPF, RBC count from 8 HPF equal 2000 RBC, Use actual RBCs/µl blood to calculate parasite density by using the following formula: parasites/µl= # of parasites in 8HPF/2000)× actual RBC.

SECONDARY OUTCOMES:
Number of participants with adverse events | vital signs: Days 1 through 6; ECG: Days1, 2, 3; Labs: Days 2, 3, 5, study completion
  Number of participants with adverse events determined by Vital sign(body temperature, blood pressure and pulse rate): pre dose, 4, 8, 12, 16, 20, 24 hours post dose on Day 1: then 6, 12, 18, 24 hours post dose on each day during domiciles period until at least two consecutive normal temperature readings are obtained, then it will measure daily until Day 6. ECG: 3-4 hours post dose on day1; pre dose, 3-4 hours post dose on Day 2; pre dose, 3-4 hours post dose on Day 3 and study completion. Lab evaluation: Day 2, Day3 and Day5, study completion.
Area under the curve (AUC)0-24h on Day 1 and Day 3 | Day 1 and Day 3
  The parent drug in plasma samples will be analyzed. On Day 1: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose. *The 24h sampling of first post dose should be taken before the second dose.
  On Day 3: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, and 192 hours post dose
The accumulation ratio (Racc) (=AUC0-24h, day3/AUC0-24h, day1) | Day 1 and Day 3
  The parent drug in plasma samples will be analyzed. On Day 1: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose. *The 24h sampling of first post dose should be taken before the second dose.
  On Day 3: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, and 192 hours post dose
Maximum concentration (Cmax) on Day 1 and Day 3 | Day 1 and Day 3
  The parent drug in plasma samples will be analyzed. On Day 1: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose. *The 24h sampling of first post dose should be taken before the second dose.
  On Day 3: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, and 192 hours post dose
Time to maximum concentration (Tmax) on Day 1 and Day 3 | Day 1 and Day 3
  The parent drug in plasma samples will be analyzed. On Day 1: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose. *The 24h sampling of first post dose should be taken before the second dose.
  On Day 3: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, and 192 hours post dose
Half-life (T1/2) | Day 3
  The parent drug in plasma samples will be analyzed On Day 3: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, and 192 hours post dose
Clearance (CL/F ) | Day 3
  The parent drug in plasma samples will be analyzed On Day 3: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, and 192 hours post dose
The apparent volume of distribution during the terminal elimination phase following extravascular administration (Vz/F) | Day 3
  The parent drug in plasma samples will be analyzed. On Day 3: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 144, and 192 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Thailand (3):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Tak
  - Novartis Investigative Site, Tak Province

REFERENCES:
- [Derived] White NJ, Pukrittayakamee S, Phyo AP, Rueangweerayut R, Nosten F, Jittamala P, Jeeyapant A, Jain JP, Lefevre G, Li R, Magnusson B, Diagana TT, Leong FJ. Spiroindolone KAE609 for falciparum and vivax malaria. N Engl J Med. 2014 Jul 31;371(5):403-10. doi: 10.1056/NEJMoa1315860. PMID 25075833